CLINICAL TRIAL: NCT06832579
Title: Pilot Study for SmartWatch-driven AF Detection in Stroke Patients
Brief Title: SmartWatch-driven AF Detection in Stroke Patients
Acronym: Find-AF2 Watch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Rolf Wachter, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Find-AF2 Watch
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Ischemic Stroke; ECG Monitoring; Secondary Prevention; Wearables
Keywords: ECG monitoring; ICM; Wearables; Stroke; ischemic stroke; atrial fibrillation; secondary prevention
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Stroke | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, multicenter interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AppleWatch (Experimental): semi-continuous heart rhythm monitoring with AppleWatch
  for 12 weeks
  Interventions: Device: Wearable
- PulseOn (Experimental): semi-continuous heart rhythm monitoring with PulseOn device
  for 12 weeks
  Interventions: Device: Wearable

INTERVENTIONS:
Device: Wearable — semi-continuous heart rhythm monitoring with Wearable

SUMMARY:
Unrecognized atrial fibrillation (AF) is a common cause of ischemic stroke. Implantable event monitors (ICM) are the gold standard for continuous heart rhythm monitoring but they have been implemented in very few patients after stroke due to high invasiveness and high costs.

In this trial, patients with implanted ICMs (Medtronic Reveal LINQ Insertable Cardiac Monitor) will be randomized to use one of two wearables (1:1 Apple Watch or PulseOn) for continuous monitoring. The aim is to compare the probability of detecting an episode of AF with a wearable versus the gold standard ICM.

Both groups will use the wearable for 12 weeks. If the wearables detect an arrhythmic pulse curve, this is communicated by vibration. By laying the other hand on the device, a 1-channel ECG is performed. ECG data will be transferred regularly to the CoreLab (Universityhospital Leipzig) for analysis.

After 12 weeks, the patients will visit the site and answer questions regarding the usability, compliance and satisfaction with the wearables.

DETAILED DESCRIPTION:
Patients with established continuous ICM monitoring from the prospective, randomized, multicenter study Find-AF 2 (NCT04371055) are recruited for this trial. Find-AF 2 is being carried out at Leipzig University Hospital since 2020 with the help of about 50 study centers throughout Germany.

The AppleWatch Series 10, a device from the current market leader, was chosen because extensive data from clinical trials is already available and data regarding the market leader has particular societal relevance. The AF detection algorithm is based on photoplethysmography (analysis of the pulse current curve) and semicontinuous monitoring. If a rhythm irregularity is detected during hourly measurements, the measurement interval is shortened. If this finding is confirmed in several consecutive measurements, the user is notified. In this pilot study, patients are trained to record a 30-second ECG with the AppleWatch in the event of notification. This is done by placing the other hand on the crown of the watch. The report will then be transmitted. The AppleWatch must be paired with another Apple device (e.g. iPhone) to use the ECG app and must be charged daily (battery life 18 hours). Our patients are provided with an iPhone for study use and are trained in using the AppleWatch.

The AppleWatch is not certified as medical device, but the ECG data collected by the AppleWatch will be used for research purposes only and not for therapeutical or diagnostical purposes.

The second wearable will be the PulseOn device. The battery lasts over two weeks. No additional device is needed for writing an ECG. AF screening is also performed photoplethysmographically. In the case of detection of an arrhythmic pulse curve, this is communicated by vibration. By laying the other hand on the device, a 1-channel ECG is performed for registration. Regular data transfer is done at the patient's home via a gateway device to the PulseOn server. The Core lab will monitor the data transmission. Although PulseOn is a certified medical device, the ECG data collected by the PulseOn device will be used for research purposes only and not for therapeutical or diagnostical purposes. The ICM is the gold standard for recording relevant arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Study participation in Find-AF 2
* Randomization in the intervention arm of the Find-AF 2 study and presence of an implanted event recorder (Medtronic Reveal LINQTM Insertable Cardiac Monitor)
* Signed informed consent
* All inclusion criteria of the Find-AF 2 study are met (according to protocol version Final 4.0, dated 08.05.2024):

  i. Recent symptomatic ischemic stroke within the last 30 days (sudden focal neurologic deficit lasting > 24 h consistent with the territory of a cerebral artery) If the neurologic deficit lasted < 24 h a corresponding lesion* on brain imaging is needed.

ii. Age ≥ 60 years. iii. Patient without or with only slight disability (modified Rankin Scale score ≤ 2) before onset of stroke-related symtoms.

iv. Written informed consent

* Corresponding lesion can be an acute lesion on diffusion-weighted magnetic resonance imaging, native computed tomography (CT) or CT perfusion imaging or a recent occlusion or intracranial thrombus on angiography (CTA, MRA, DSA)

Exclusion Criteria:

* Expiration of the battery of the event recorder in <3 months
* No in ICM data transmission possible (e. g. missing compliance)
* Poor ECG data quality according to core lab evaluation (e.g. permanent oversensing), which prevents meaningful evaluation of the event recorder data
* Exclusion criteria of the Find-AF 2 study (according to protocol version Final 4.0, dated 08.05.2024):

  i. Known history of atrial fibrillation/flutter or atrial fibrillation/flutter on admission ECG.

ii. Current indication or contraindication for oral anticoagulation at randomisation.

iii. Intracerebral bleeding in medical history iv. Patient scheduled for ECG-monitoring lasting > 7 days (Holter-ECG, implanted loop recorder, etc.).

v. Implanted pacemaker device or cardioverter/defibrillator or implanted cardiac monitor.

vi. Patient not willing to be treated with oral anticoagulants vii. Carotid artery stenosis ipsilateral to the current ischemic stroke needing operation or intervention.

viii. History of carotid endarterectomy or percutaneous stent intervention of cerebral or cervical artery within the last 30 days.

ix. Life expectancy <1 year for reasons other than stroke (e.g. metastatic cancer).

x. Patients under legal supervision or guardianship xi. Psychological/mental or other inabilities to supply required information (e.g. fill out the questionnaire due to dementia, language difficulties, ... ) or participate in the required tests xii. Participation in other randomized interventional trials xiii. Suspected lack of compliance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
sensitivity as a function of AF duration | from the date of device handover to the date of device return
  the probability that an AF episode will be detected as it depends on the duration of the episode

SECONDARY OUTCOMES:
Time worn | from the date of device handover to the date of device return
  the proportion of time that the wearable collected and transferred data
Detection sensitivity as a function of AF duration | from the date of device handover to the date of device return
  If the device is being worn during at least 120 seconds of an AF episode, what is the probability of its informing the patient of an arrhythmia?
ECG compliance | from the date of device handover to the date of device return
  if the wearable informs of an episode, what is the probability that the patient will let the device save an ECG
Overall sensitivity | from the date of device handover to the date of device return
  For patients who had at least one AF episode, what is the probability that the wearable claims there was at least one episode?
Time to first ECG-confirmed AF episode | from the date of device handover to the date of device return
Overall specificity | from the date of device handover to the date of device return
  for patients who had no AF episodes, what is the probability that there is no ECG confirmation of any episodes?
False discovery rate (1-PPV (positive predictive value) | from the date of device handover to the date of device return
  For every ECG-confirmed episode found by the wearable, the gold standard episode definition will be used for comparison
For the ICM: What proportion of detected signals are available as ECGs? | from the date of device handover to the date of device return
For the ICM: What is the false discovery rate of the available ECGs? | from the date of device handover to the date of device return
Do patients with an ICM claim to be willing to be randomized to an ICM vs a wearable? | after 12 weeks
Patient satisfaction with the wearable | after 12 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (13):
  - RHÖN-KLINIKUM Campus Bad Neustadt Von-Guttenberg-Straße 11 Akutneurologie II - Stroke Unit - klinische Forschung, Bad Neustadt an der Saale
  - Evangelisches Klinikum Bethel, Clinic for Neurology, Bielefeld
  - Medizinische Fakultät Carl Gustav Carus Klinik und Poliklinik für Neurologie, Dresden
  - University of Essen, Clinic of Neurology, Essen
  - University of Göttingen, Clinic for Neurology, Göttingen
  - Bezirkskrankenhaus Günzburg Klinik für Neurologie und Neurologische Rehabilitation Ludwig-Heilmeyer-Straße 2, Günzburg
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Klinik für Neurologie Klinikum Ibbenbüren Große Str. 41, Ibbenbueren
  - University Hospital Leipzig, Clinic for Neurology, Leipzig
  - University of Mainz, Clinic for Neurology, Mainz
  - Johannes Wesling Klinikum Minden Universitätsklinik für Neurologie und Neurogeriatrie Hans-Nolte-Str. 1, Minden
  - Klinik für Neurologie Universitätsklinik der Paracelsus Medizinischen Privatuniversität Breslauer Str. 201, Nuremberg
  - Kliniken Südostbayern AG, Klinikum Traunstein, Traunstein

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication of the major results